CLINICAL TRIAL: NCT00796809
Title: Risk of Coccidioidomycosis in Patients Receiving Anti-TNF and Other Biologic Agents for an Inflammatory Arthritis
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-0930-04
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Coccidioidomycosis; Rheumatoid Arthritis
Keywords: TNF inhibitors; Biologic agents; coccidioidomycosis; Rheumatoid arthritis
MeSH Terms: conditions — Coccidioidomycosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Biologics: Patients receiving TNF inhibitors or biologic agents
- DMARD: Patients receiving methotrexate without any biologic

SUMMARY:
The goal of the project is to study the risk of coccidioidomycosis (valley fever) in patients receiving anti-TNF and other biologic agents for inflammatory arthritis in Tucson, Arizona.

DETAILED DESCRIPTION:
Retrospective chart review of all patients with an inflammatory arthritis seen at the University Rheumatology clinic since January 2000.

ELIGIBILITY:
Inclusion Criteria:

* All active patients with an inflammatory arthritis seen at the University of Arizona from January 2000

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an inflammatory arthritis receiving care at our Rheumatology ambulatory clinic at the University of Arizona
Sampling Method: Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Determine the incidence rate and calculate the risk of coccidioidomycosis in patients receiving various anti-TNF agents or other biologics, and patients not receiving these agents for their inflammatory arthritis | one year

SECONDARY OUTCOMES:
To calculate the incidence density of coccidioidomycosis cases in patients receiving each drug. | One year
To compare number of disseminated cases of coccidioidomycosis in each group | One year

CONTACTS AND LOCATIONS:
Overall Officials: Berchman A Vaz, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona - Arizona Arthritis Center, Tucson, Arizona, United States